CLINICAL TRIAL: NCT00524238
Title: Impact of Hypothyroidism on Glucose, Lipid, and Amino Acid Turnover
Brief Title: Metabolic Changes in Hypothyroid Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Signe Gjedde, MD, Medical Department M, Aarhus Sygehus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20030196
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-02

CONDITIONS: Hypothyroidism
Keywords: hypothyroidism; glucose turnover; clamp; insulin resistance; lipid turnover; amino acid turnover
MeSH Terms: conditions — Hypothyroidism; Insulin Resistance | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): 11 hypothyroid patients, newly diagnosed, examined before and after treatment
  Interventions: Drug: L-thyroxine
- 2 (No Intervention): 10 healthy controls

INTERVENTIONS:
Drug: L-thyroxine — The hypothyroid patients receive usual treatment with L-thyroxine in our out patient clinic. The doctors there subscribe the medication, this study has no protocol regarding this, we observe the patients again after having been biochemically euthyroid for at least two months.
  Arms: 1

SUMMARY:
Hypothyroidism is a frequent condition in danish women, but often overlooked. Along with fatigue one of the main symptoms is weight gain as a result to significantly decreased energy expenditure.

This study was undertaken to elucidate changes in glucose, lipid and amino acid turnover in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed hypothyroidism with tsh over 40 mU/L, etiology chronic autoimmune thyroiditis
* Healthy controls matched regarding sex, age and body mass index

Exclusion Criteria:

* Pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Signe Gjedde, MD, Principal Investigator — Aarhus University, Clinical Institute
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Gjedde S, Gormsen LC, Riis AL, Jorgensen JO, Rungby J, Moller N, Weeke J, Pedersen SB. Reduced expression of uncoupling protein 2 in adipose tissue in patients with hypothyroidism. J Clin Endocrinol Metab. 2010 Jul;95(7):3537-41. doi: 10.1210/jc.2009-0907. Epub 2010 Apr 28. PMID 20427509